CLINICAL TRIAL: NCT00002217
Title: Combivir, 1592U89, 141W94 Triple Antiretroviral, Experienced Patient Trial
Brief Title: A Study of Combivir Plus Abacavir Plus 141W94 in Patients Who Previously Have Used Anti-HIV Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 280D; UNAP 12; NZTA 4005
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-05

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Patient Compliance; Anti-HIV Agents; abacavir
MeSH Terms: conditions — HIV Infections; Patient Compliance | interventions — lamivudine, zidovudine drug combination; abacavir; amprenavir

INTERVENTIONS:
Drug: Lamivudine/Zidovudine
Drug: Abacavir sulfate
Drug: Amprenavir

SUMMARY:
The purpose of this study is to test the effectiveness of Combivir plus abacavir plus 141W94 in patients who previously have used anti-HIV drugs.

DETAILED DESCRIPTION:
In this open-label study antiretroviral-experienced patients receive Combivir (3TC/AZT tablet) plus 1592U89 (abacavir) and 141W94 twice daily for 48 weeks.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* CD4 count greater than 50 cells/mm3.
* HIV RNA less than 50,000 copies/ml.
* No active AIDS (excluding CD4 count less than 200 cells/mm3).
* Ability to comply with dosing schedule and protocol evaluations.

Prior Medication:

Allowed:

AZT or non-nucleoside reverse transcriptase inhibitors (NNRTIs).

Exclusion Criteria

Co-existing Condition:

Patients with any of the following symptoms or conditions are excluded:

* Active AIDS (not excluding CD4 count less than 200).
* Malabsorption syndrome affecting drug absorption.
* Serious medical condition that would compromise safety of the patient.

Concurrent Medication:

Excluded:

* AZT or NNRTIs.
* More than 1 week treatment with any protease inhibitor.
* Enrollment in any other investigational drug protocol.

Patients with the following prior conditions are excluded:

History of clinically relevant pancreatitis or hepatitis within the past 6 months.

Required:

Antiretroviral therapy with either single or double reverse transcriptase inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Anderson Clinical Research, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Henry K, Shaeffer M, Ross L, Johnson M, Fisher R, Liao Q, Graham N. Response to Combivir and abacavir given bid to nucleoside experienced patients is not affected by the presence of the M184V mutation. 6th Conf Retro and Opportun Infect. 1999 Jan 31 - Feb 4 (abstract no 132)
- [Background] Henry K, Wallace RJ, Bellman PC, Norris D, Fisher RL, Ross LL, Liao Q, Shaefer MS; TARGET Study Team. Twice-daily triple nucleoside intensification treatment with lamivudine-zidovudine plus abacavir sustains suppression of human immunodeficiency virus type 1: results of the TARGET Study. J Infect Dis. 2001 Feb 15;183(4):571-8. doi: 10.1086/318527. Epub 2001 Jan 11. PMID 11170982